CLINICAL TRIAL: NCT01166360
Title: The Prognostic Relevance of Cerebral Oxygen Saturation, NTproBNP and Preoperative Creatinine Clearance in Cardiac Surgical Patients; Amendment 4: the Prognostic Relevance of Growth Differentiation Factor 15 (GDF-15) and High Sensitive Troponin-t (hsTnT)
Brief Title: The Usefulness of Growth Differentiation Factor 15 (GDF-15) for Risk Stratification in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Prof. Dr. med. Matthias Heringlake, Department of Anesthesiology, University of Luebeck
Other Study IDs: CS_RS_2008-2009 - GDF_TNT
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Heart Failure; Coronary Artery Disease
Keywords: Risk prediction; Euroscore; GDF-15; hsTnT; cardiac surgery
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients 2009: Patients undergoing cardiac surgery in 2009
- Patients 2008: Patients undergoing cardiac surgery in 2008

SUMMARY:
Growth determination factor 15 (GDF-15) and high sensitive troponin-t (hsTnT) are emerging humoral markers for risk stratification in clinically stable heart failure patients and in patients with stable coronary artery disease. No data are available about the prognostic value of these peptides in relation to mortality and morbidity in patients undergoing cardiac surgery.

Primary objective of the present study is to test the hypothesis, that GDF-15 is superior to a standard preoperative risk score, the additive Euroscore for the prediction of 30 day mortality and postoperative morbidity in patients scheduled for cardiac surgery.

Secondary objectives are to test the predictive value of hsTNT, either alone, or in combination with GDF-15 and if GDF-15 adds additional information to NTproBNP levels and preoperative cerebral oxygen saturation (ScO2) levels.

DETAILED DESCRIPTION:
The study will be based on 2 patient cohorts, a group of patients studied during an observation period (2009) and a validation cohort of patients studied in 2008. The 2009 cohort (about 800 patients) will be analyzed to determine the predictive value of GDF-15 for predicting mortality and morbidity. The 2008 cohort (about 1200 patients) will be used to validate these findings.

Besides conventional morbidity markers, new sensitive markers of organ dysfunction (FABP, NGAL, sFLT-1, PIGF) will also be tested in the 2009 group.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cardiac surgery

Exclusion Criteria:

* Withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing primary cardiac surgery at a University hospital.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
30 day mortality | 30 days
  The predictive accuracy of GDF-15 will be compared with the Euroscore. Since the Euroscore has been calibrated for 30 day mortality, this time frame will be used as primary outcome parameter.

SECONDARY OUTCOMES:
1 year mortality | 365 days
  1 year mortality is a more relevant outcome variable than 30 day mortality
Renal dysfunction defined according to AKI-criteria | 30 days
  Renal dysfunction is an important outcome variable in cardiac surgery.
MaC score as combined measure of postoperative morbidity | 30 days
  The MACS is a combined score for postoperative complications: low cardiac output syndrome, need for renal replacement therapy, stroke, reintubation.
Sensitive markers of organ dysfunction | 4 days
  Fatty acid binding protein, neutrophyil gelatinase associated lipocalin are sensitive markers of organ dysfunction and shall be used to give more precise information on organ dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Heringlake, MD, Principal Investigator — Department of Anesthesiology, University of Luebeck
Locations (1):
- Department of Anesthesiology, University of Luebeck, Lübeck, Germany

REFERENCES:
- [Derived] Heringlake M, Charitos EI, Erber K, Berggreen AE, Heinze H, Paarmann H. Preoperative plasma growth-differentiation factor-15 for prediction of acute kidney injury in patients undergoing cardiac surgery. Crit Care. 2016 Oct 8;20(1):317. doi: 10.1186/s13054-016-1482-3. PMID 27717384
- [Derived] Heringlake M, Charitos EI, Gatz N, Kabler JH, Beilharz A, Holz D, Schon J, Paarmann H, Petersen M, Hanke T. Growth differentiation factor 15: a novel risk marker adjunct to the EuroSCORE for risk stratification in cardiac surgery patients. J Am Coll Cardiol. 2013 Feb 12;61(6):672-81. doi: 10.1016/j.jacc.2012.09.059. PMID 23391200